CLINICAL TRIAL: NCT06892912
Title: Multicenter Prospective Observational Study on Diaphragmatic Function Assessment by Ultrasound in Patients with Acute Respiratory Failure Receiving Non-invasive Mechanical Ventilation or High Flow Nasal Canula
Acronym: DIAFUSION
Status: Not yet recruiting | Type: Observational
Sponsor: Foro Internacional en Cuidado Crítico (Other)
Responsible Party: Principal Investigator, Carlos Andres Santacruz Herrera, Principal investigator, Foro Internacional en Cuidado Crítico
Other Study IDs: CBE03_2025
Record Dates: First submitted 2025-03-14; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Respiration Disorders
Keywords: Respiratory failure; Diaphragmatic ultrasound; Respiratory support
MeSH Terms: conditions — Respiration Disorders; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with acute respiratory failure: Patients with acute respiratory failure (e.g., hypoxemic or hypercapnic) who require non-invasive mechanical ventilation or high-flow nasal canula.
  Interventions: Other: Diaphragmatic ultrasound

INTERVENTIONS:
Other: Diaphragmatic ultrasound — Sample:
  Given the observational nature of the study, a convenience sample will be obtained from all patients admitted to the emergency services and/or ICU with respiratory failure over the course of 1 year.
  Inclusion Criteria:
  * Age ≥ 18 years
  * Hypoxemic respiratory failure (SpO2 < 88% - PaO2 < 60 mmHg) or hypercapnic (PaCO2 > 40)
  * Need for NIMV and/or HFNC.
  Exclusion Criteria:
  * Neuromuscular disease
  * Pregnancy
  * Tracheostomy
  * Rib fractures
  * Cervical injuries
  * Diaphragmatic paralysis
  * Diaphragmatic malformations
  * Hemodynamic instability
  * Morbid obesity (BMI > 35)
  * Use of sedation and neuromuscular relaxants
  * Pneumothorax or pneumomediastinum
  * Poor acoustic window
  * Critically ill patients with a prognosis of less than 24 hours of life
  * Patients receiving palliative interventions.

SUMMARY:
The primary goal of this study is to assess diaphragm function in patients with acute respiratory failure before and during the use of high-flow oxygen and/or non-invasive breathing support. The key question it seeks to answer is:

1. How do ultrasound measurements of diaphragmatic function vary with different levels of breathing support in patients with acute respiratory failure? Participants with acute respiratory failure will undergo diaphragmatic ultrasound evaluation as part of their standard medical care at various levels of respiratory support.

DETAILED DESCRIPTION:
Protocol for Assessment and Measurement of Diaphragmatic Ultrasound

Ultrasonographic Evaluation of the Diaphragm Protocol:

This protocol focuses on observing and evaluating diaphragmatic function in patients with acute respiratory failure who require non-invasive mechanical ventilation (NIMV) and/or high-flow nasal cannula (HFNC). The ultrasound measurements performed by researchers will be standardized to ensure consistency and accuracy in assessing diaphragmatic function.

Assessment of Diaphragmatic Thickness Collection of arterial blood gases is performed 1 hour after being on the clinician-selected pressure support (PS) level.

Cut-Off Points for Diaphragmatic Assessment Parameters

For the evaluation of diaphragmatic function in patients with acute respiratory failure requiring non-invasive mechanical ventilation (NIMV), the following cut-off points will be used:

Diaphragmatic Excursion:

Diaphragmatic excursion will be measured in centimeters using ultrasound in B-mode and M-mode.

Cut-Off Point: A diaphragmatic excursion of less than 1 cm will be considered indicative of severe diaphragmatic dysfunction, while an excursion greater than 2 cm will be interpreted as excessive diaphragmatic function.

Time to Maximum Inspiratory Amplitude:

This parameter will be measured in seconds from the start of inspiration until the diaphragm reaches its maximum amplitude.

Cut-Off Point: A time to maximum amplitude greater than 0.5 seconds will suggest compromised diaphragmatic function, while a time of less than 0.5 seconds will be deemed normal.

Diaphragmatic Thickening Fraction:

To evaluate diaphragmatic thickness, the following methodology will be implemented:

Patient Positioning:

Explain the procedure to the patient and/or family member. The patient should be positioned supine with the head of the bed elevated between 30 and 40 degrees.

Equipment Setup:

Select a high-frequency linear transducer (7-10 Megahertz) in B-mode. Position the probe in the right intercostal space, drawing an imaginary line between the anterior axillary line and the mid-axillary line, between the eighth and tenth right ribs.

The transducer must be positioned consistently in the same location for each measurement.

Identification of the Apposition Zone:

Locate the apposition zone of the diaphragm, which will appear as a three-layered structure: a central non-echoic layer (the diaphragm) surrounded by two parallel echogenic layers (the peritoneum and the diaphragmatic pleura).

Measurement of Thickness:

In M-mode, the thickness of the diaphragm will be evaluated, which varies according to the phase of the respiratory cycle, being greater during inspiration and less during expiration.

The sweep speed will be increased to obtain at least three consecutive thickening measurements on the screen. The image will be frozen, and three measurements will be taken during three different breaths to obtain an average.

During inspiration, it will be ensured that the thickness is greater, and the distance between the hyperechoic lines will be measured.

During expiration, the distance between the hyperechoic lines will be measured, ensuring that the thickness is less.

Measurement of Diaphragmatic Excursion:

To evaluate diaphragmatic excursion, the following methodology will be implemented:

Patient Positioning:

Explain the procedure to the patient and/or family member. The patient should be positioned supine with the head of the bed elevated between 30 and 40 degrees.

Equipment Setup:

A sector transducer (5-8 Megahertz) or a convex transducer (2-5 Megahertz) will be used in B-mode.

The probe will be positioned in the mid-clavicular line window, immediately below the costal margin, between the mid-clavicular line and the anterior axillary line. The ultrasound beam will be directed cephalically, perpendicular to the posterior third of the diaphragm.

The transducer must be positioned consistently in the same location for each measurement.

Ultrasound of the Diaphragmatic Dome Area:

Using a sector transducer in a cephalic position, the diaphragm will be insonated, adjusting the image so that M-mode is at a 90-degree angle to the dome of the diaphragm.

The sweep speed will be increased to obtain at least three consecutive excursions displayed on the screen. The image will be frozen, and three measurements will be taken during three different breaths to obtain an average.

Measurements of Diaphragmatic Function by Ultrasound

Calculation of Diaphragmatic Thickening Fraction:

This will be calculated by taking the thickening diameter during inspiration, subtracting the thickening diameter during expiration, dividing the result by the thickening diameter during expiration, and multiplying the result by 100%. The diaphragmatic thickening fraction, which varies depending on ventilation support, has reference values indicating diaphragmatic insufficiency (less than 20%) and values above 30%.

Calculation of Diaphragmatic Excursion:

Diaphragmatic excursion (DE, centimeters), inspiratory time (TPIA-dia, seconds), diaphragm contraction speed (DE/TPIA-dia, centimeters per second), and total time (Ttot, seconds) will be calculated in M-mode; diaphragmatic dysfunction will be defined as DE < 1 cm or paradoxical movement.

Record the data in the corresponding format. Conduct the measurements at the selected flow levels of the high-flow nasal cannula.

The thickening fraction will be calculated using the formula:

((\text{Thickness during Inspiration} - \text{Thickness during Expiration}) / \text{Thickness during Expiration} \times 100%) Cut-Off Point: A thickening fraction of less than 20% will be considered indicative of diaphragmatic weakness, while a fraction greater than 30% will be deemed excessive.

These cut-off points will allow for a precise and objective assessment of diaphragmatic function, facilitating optimal titration of support pressure during non-invasive mechanical ventilation (NIMV) and thereby improving clinical outcomes in patients with acute respiratory failure.

Study Protocol:

The protocol begins with the admission of the patient with hypoxemic/hypercapnic respiratory failure. Support pressure levels (NIMV cohort) / flow (high-flow nasal cannula (HFNC) cohort) will be applied at the discretion of each center. Patients will be placed in a semi-sitting position at an angle of 30-40 degrees throughout the study. The first diaphragmatic measurement will be taken before the initiation of non-invasive mechanical ventilation (T0) without delaying the start of treatment. The second measurement will be taken 30 minutes after the start of NIMV/HFNC (T1), and the third will be taken 60 minutes after the start of NIMV/HFNC (T2). Measurements will include excursion (centimeters), time to maximum inspiratory amplitude (seconds), total respiratory cycle time (seconds), and diaphragmatic thickening fraction (ED, centimeters) (FTD%), as well as oxygen saturation (SpO2), exhaled tidal volume, respiratory rate, heart rate, and systolic, diastolic, and mean blood pressure at each time point (T0, T1, and T2).

The next measurement of hemodynamic variables (systolic, diastolic, mean blood pressure, heart rate) and respiratory variables (respiratory rate, SpO2) will be conducted one hour after identifying the optimal level of support pressure/flow (defined individually by each center) at which the patient will remain.

Summary of Ultrasonographic Diaphragm Assessment:

Non-Invasive Mechanical Ventilation (NIMV) Patient Cohort Time 0: Prior to the initiation of NIMV support. Time 1: 30 minutes after the initiation of NIMV. Time 2: 60 minutes after the initiation of NIMV.

High-Flow Nasal Cannula (HFNC) Patient Cohort Time 0: Prior to the initiation of HFNC support. Time 1: 30 minutes after the initiation of HFNC. Time 2: 60 minutes after the initiation of HFNC.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Hypoxemic respiratory failure (SpO2 < 88% - PaO2 < 60 mmHg) or hypercapnic (PaCO2 > 40)
* Need for NIMV and/or HFNC.

Exclusion Criteria:

* Neuromuscular disease
* Pregnancy
* Tracheostomy
* Rib fractures
* Cervical injuries
* Diaphragmatic paralysis
* Diaphragmatic malformations
* Hemodynamic instability
* Morbid obesity (BMI > 35)
* Use of sedation and neuromuscular relaxants
* Pneumothorax or pneumomediastinum
* Poor acoustic window
* Critically ill patients with a prognosis of less than 24 hours of life Patients receiving palliative interventions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute respiratory failure in the emergency department or intensive care unit (ICU).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06-02 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Correlation of Diaphragmatic Function (Excursion and Thickening Fraction) with Ventilatory Support Effectiveness in Patients with Acute Respiratory Failure | From enrollment to ICU discharge (aprox. 2 weeks)
  To evaluate the relationship between diaphragmatic function measured by ultrasound (excursion and thickening fraction) prior to and during the administration of non-invasive respiratory support. This evaluation will focus on the effectiveness of ventilatory support in terms of improvement in respiratory mechanics parameters and the reduction in the need for orotracheal intubation in patients with acute respiratory failure (hypoxemic/hypercapnic).

SECONDARY OUTCOMES:
Correlation of Diaphragmatic Function (Excursion and Thickening Fraction) with Respiratory Mechanics, Ventilation Duration, and ICU Mortality in Patients with Acute Respiratory Failure | From enrollment to ICU discharge (aprox. 2 weeks)
  Evaluate the relationship between diaphragmatic excursion (cm), time to maximum inspiratory amplitude (s), total respiratory cycle time (s), and diaphragmatic thickening fraction (%) during titration of support pressure (NIMV) or flow (HFNC) with variables such as exhaled tidal volume (ml), respiratory rate (breaths/min), oxygen saturation (SpO2 %), arterial blood gases (PaO2/FiO2 ratio, PaCO2), arterial lactate (mmol/L), heart rate (beats/min), and blood pressure (mmHg).
  Analyze differences in diaphragmatic excursion (cm) and parameters between patient subgroups based on oxygenation (hypoxemic vs. hypercapnic) and infection status (septic vs. non-septic).
  Investigate correlations between diaphragmatic excursion (cm) and thickening fraction (%) with ICU length of stay.
  Assess relationships between diaphragmatic function (excursion cm, thickening fraction %) and days on NIMV and invasive ventilation.
  Determine correlations between diaphragmatic function (excursion cm, thickening frac

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Santacruz H, MD, PhD, Study Director — Foro Internacional en Cuidado Crítico

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.